CLINICAL TRIAL: NCT01149447
Title: Prospective Clinical Follow-up of Patients Presenting With Cryptogenic Stroke Treated With the Percutaneous Closure of a Patent Foramen Ovale
Brief Title: Prospective Clinical Follow-up After the Percutaneous Closure of a Patent Foramen Ovale
Acronym: PFO-HUG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Robert F Bonvini, MD, University Hospital, Geneva
Other Study IDs: PFO-HUG-Study
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Stroke; Foramen Ovale, Patent
Keywords: cryptogenic stroke; percutaneous closure of PFO; follow-up exams
MeSH Terms: conditions — Stroke; Foramen Ovale, Patent; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Following a cryptogenic stroke, many patients are nowadays treated with the percutaneous closure of a patent foramen ovale (PFO), assuming that the aetiology of the stroke is secondary to a paradoxical embolism. After the PFO closure procedure a dual antiplatelet regimen is often prescribed for 3-6 months and several cardiologic and neurologic follow-up exams are scheduled in the first 12 months of follow-up. Usually a transthoracic +/- transoesophageal echocardiography (TTE +/- TEE) are performed at 6 months, however this kind of control is not systematically performed. In order to improve the clinical outcomes in this young patients' population, the investigators prospectively perform a complete cardiologic and neurologic follow-up program to all patients undergoing a successful percutaneous closure of a PFO.

The aim of these controls is to confirm the good position of the PFO-device, to confirm the absence of any residual right to left shunt or any significant atrial arrhythmias Furthermore this prospective follow-up will analyze the possible mechanisms leading to a cerebral stroke recurrence (e.g. size of the PFO, presence of an atrial septal aneurysm, presence of a residual shunt, size of the utilized closure device, ....).

DETAILED DESCRIPTION:
At follow-up the following exams will be performed:

* at hospital discharge: chest X-ray +/- TTE + 7-days event loop record (ELR)
* at 6 months: clinical cardiologic and neurologic examination + TTE + TEE + 7-days ELR + trans-cranial doppler (TCD) with micro bubbles detection.
* at 1 year: clinical cardiologic and neurologic examination + TTE +/- TEE + 7-days ELR + trans-cranial doppler (TCD) with micro bubbles detection +/- cerebral MRI

ELIGIBILITY:
Inclusion Criteria:

* 18 years old patients
* signed informed consent
* all consecutive patients undergoing a successful percutaneous closure of a PFO secondary to a cryptogenic stroke

Exclusion Criteria:

* all patients with an alternative aetiology of the initial stroke
* all patients in whom the percutaneous closure of the PFO is contraindicated
* all patients with a known allergy to aspirin and or clopidogrel

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all consecutive patients presenting with a cryptogenic stroke, in whom a successful percutaneous closure of their PFO is performed
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2001-01

PRIMARY OUTCOMES:
residual shunt at 6-12 months follow-up | 6-12 months
  incidence and clinical relevance of right to left residual shunts at 6-12 months after the successful closure of the PFO
stroke recurrence | 6-12 months
  incidence and clinical predictors of stroke recurrence at 6-12 months
possible other aetiologies of the initial cryptogenic stroke | 6-12 months
  during the 12 months follow-up all other possible aetiologies explaining the initial cryptogenic stroke will be taken into consideration

SECONDARY OUTCOMES:
6 months dual antiplatelet regimen safety and efficacy | 6 months
  confirm the safety and efficacy of the adopted 6 months dual antiplatelet regimen

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Bonvini, MD, Principal Investigator — University of Geneva
Locations (1):
- University of Geneva, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- See also: university of geneva web site — http://www.hug-ge.ch